CLINICAL TRIAL: NCT00147108
Title: Phase 3 Study of MR Guided Focused Ultrasound Surgery in the Treatment of Breast Fibroadenomas
Brief Title: MR Guided Focused Ultrasound Surgery in the Treatment of Breast Fibroadenomas
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BF002
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-09

CONDITIONS: Breast Fibroadenoma
Keywords: Breast Cancer
MeSH Terms: conditions — Fibroadenoma; Breast Neoplasms

INTERVENTIONS:
Device: ExAblate 2000

SUMMARY:
The primary objective of this pivotal study is to evaluate the safety and efficacy of FUS treatment of breast fibroadenomas. Our hypothesis is that FUS lesion ablation of a fibroadenoma will have the following results: a. lead to a decrease in lesion cross-sectional area of > 50% on palpation, and >65% in lesion volume as measured by MRI (both calculations assume an elliptical shape of the lesion in all 3 dimensions). b. this decrease in size, along with the softening of the treated volume will result in satisfactory clinical results in greater than 50 % of the patients.

DETAILED DESCRIPTION:
Many patients are now diagnosed with breast fibroadenomas. These are generally detected during breast self-exams, or annual physicals as a smooth, rubbery, oval/elliptical lump in the breast. These patients then go on to receive mammograms, sonograms and usually a core biopsy for the differential diagnosis of benign disease (fibroadenoma) vs breast cancer. Although fibroadenomas are benign, they can be of great concern to the patient because of their ability to mask the presence of other lumps in the breast, they can be painful, cause a physical deformity of the breast or have other symptoms. The current treatment is surgical excision. Surgical removal is invasive and may be cosmetically undesirable to some patients. It would be advantageous to develop a non-invasive ablative method for treatment of this disease. Measures of the clinical success of patients who elect surgical removal of fibroadenomas are generally subjective, and evaluated primarily by the patient (lack of palpable lesion, pain free, and an acceptable cosmetic result). A non-randomized study is proposed to allow for a more practical approach in subject recruitment. Analysis on safety and efficacy will be performed through the use of MRI evaluation and physical exams.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Females only
* Histologic confirmation of breast fibroadenoma by large core (needle gauge range 11-14 ) biopsy.
* Single tumor per breast quadrant
* Tumor clearly visible on non-contrast MRI
* Age > 18 years 3.2.6 Signed informed consent
* Tumor 5 mm or larger as measured on pre-treatment MR.

Exclusion Criteria:

* Gender: male
* Focal breast lesion on MRI over 3.5 cm as evaluated by MRI
* Distance from the edge of the breast fibroadenoma to the skin less than 0.5-cm or ribs less than 1 cm.
* Microcalcifications within the lesion
* Known intolerance to the MRI contrast agent (Gadolinium or Magnevist) 3.3.6 Patients on dialysis.
* Hemolytic anemia (hematocrit<30)
* Patients with unstable cardiac status including: Unstable angina pectoris on medication Patients with documented myocardial infarction within six months of protocol entry Congestive heart failure requiring medication (other than diuretic) Patients on anti-arrhythmic drugs Severe hypertension (diastolic BP > 100 on medication)
* Patients with cardiac pacemakers
* ASA Score>2
* Severe cerebrovascular disease (multiple CVA or CVA within 6 months) 3.3.12 Individuals who are not able or willing to tolerate the required prolonged stationary prone position during treatment (approximately 3 hrs.) 3.3.13 Patients with breast implants
* Large patients who cannot fit in the magnet (weight>250 pounds), and patients with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices
* Patients on anti-coagulation therapy, or those with an underlying bleeding disorder.
* Patient has a prior history of breast cancer
* Patient has a prior history of laser or radiation therapy to the target breast
* Patient has a prior history of chemo therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2003-01; Primary Completion 2005-08 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
treatment/ablation of breast fibroadenoma

CONTACTS AND LOCATIONS:
Overall Officials: Clare Tempany, M.D., Principal Investigator — Brigham and Women's Hospital; Robert Min, M.D., Principal Investigator — Cornell Vascular; Fred Steinberg, M.D., Principal Investigator — University MRI; Mark DeLaurentis, M.D., Principal Investigator — Virtua; Hidemi Furusawa, M.D., Principal Investigator — Breastopia Hospital
Locations (5):
- United States (4):
  - University MRI, Boca Raton, Florida
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Virtua, Voorhees Township, New Jersey
  - Cornell Vascular, New York, New York
- Breastopia Namba Hospital, Miyazaki-ken, Japan

REFERENCES:
- See also: Sponsor web page — http://www.insightec.com